CLINICAL TRIAL: NCT03952156
Title: A Phase 1/2 Open-Label, Randomized, Concurrently-Controlled, Dose Escalation Study to Evaluate the Safety and Efficacy of HMI-102 in Adult PKU Subjects With PAH Deficiency
Brief Title: Gene Therapy Clinical Study in Adult PKU
Acronym: pheNIX
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Homology Medicines has discontinued the development of this program.
Sponsor: Homology Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HMI-102-101
Record Dates: First submitted 2019-05-09; First posted 2019-05-16 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Phenylketonurias; PAH Deficiency
Keywords: PKU; Phenylketonuria; PAH Deficiency; Hyperphenylalaninemia; Phenylalanine; Adeno Associated Virus; AAVHSC15
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): Dose Level 1 of HMI-102 delivered intravenously one time
  Interventions: Genetic: HMI-102
- Cohort 2 (Experimental): Dose Level 2 of HMI-102 delivered intravenously one time
  Interventions: Genetic: HMI-102
- Cohort 3 (Experimental): Dose Level 3 of HMI-102 delivered intravenously one time
  Interventions: Genetic: HMI-102
- Delayed Treatment Control (Experimental): Delayed Treatment Control Arm
  Interventions: Genetic: HMI-102
- Expansion Phase First Dose level (Experimental): Expansion Phase First Dose Level of HMI-102 delivered intravenously one time
  Interventions: Genetic: HMI-102
- Expansion Phase Second Dose level (Experimental): Expansion Phase Second Dose Level of HMI-102 delivered intravenously one time
  Interventions: Genetic: HMI-102

INTERVENTIONS:
Genetic: HMI-102 — HMI-102 is an AAVHSC15 vector containing a functional copy of the human PAH gene
  Arms: Cohort 1; Cohort 2; Cohort 3; Expansion Phase First Dose level; Expansion Phase Second Dose level
Genetic: HMI-102 — Control subjects will generally have the same assessments as treated subjects.
  Control subjects will undergo pre-baseline procedures to confirm that they are eligible to receive treatment with HMI-102. Once eligible control subjects are dosed with HMI-102, they will initiate the same post-dose procedures as subjects who received HMI-102.
  Arms: Delayed Treatment Control

SUMMARY:
This is a Phase 1/2, open-label, randomized, concurrently-controlled, dose escalation study to evaluate the safety and efficacy of HMI-102 in adult PKU subjects with PAH deficiency. Participants will receive a single administration of HMI-102 and will be followed for safety and efficacy for 1 year.

DETAILED DESCRIPTION:
Part 1 of this study will evaluate the safety and efficacy of HMI-102 gene therapy in adult subjects with PKU due to PAH deficiency. Subjects will receive a single dose of HMI-102 administered intravenously. Up to 3 dose levels of HMI-102 may be investigated in this study. At a given dose level, a minimum of 2 subjects will be enrolled and dosed. Dosing of the first two subjects will be staggered. Following evaluation of data from the first 2 subjects in a cohort, a decision can be made to either escalate to the next dose level or expand the cohort at the selected dose level. Additional doses may be added by HMI to investigate intermediate or higher doses.

In Part 2 dose expansion, evaluation of up to 2 dose levels is planned. Subjects will be randomized to receive HMI-102 or a concurrent delayed treatment control arm. Subjects in the delayed treatment control will be eligible to receive HMI-102 after 28 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Adults 18-55 years of age at the time of informed consent
* Diagnosis of phenylketonuria (PKU) due to PAH deficiency
* Two plasma Phe values with a concentration of ≥ 600 μmol/L drawn at least 72 hours apart during the screening period and at least one historical value ≥ 600 μmol/L in the preceding 24 months.
* Subject has the ability and willingness to maintain their baseline diet, whether Phe-restricted or unrestricted for the duration of the trial, unless otherwise directed

Key Exclusion Criteria:

* Subjects with PKU that is not due to PAH deficiency
* Presence of anti-AAVHSC15 neutralizing antibodies
* ALT > ULN and AST > ULN
* Alkaline phosphatase > ULN.
* Total bilirubin > ULN, direct bilirubin > ULN
* Serum creatinine >1.5x ULN
* International normalized ratio (INR) > 1.2
* Hematology values outside of the normal range (hemoglobin <11.0 g/dL for males or <10.0 g/dL for females; white blood cells (WBC) <3,000/μL; absolute neutrophils <1500/μL; platelets <100,000/μL)
* Hemoglobin A1c >6.5% or fasting glucose >126 mg/dL
* Any clinically significant abnormal laboratory result at screening, in the opinion of the Investigator
* Contraindication to corticosteroid use or conditions that could worsen in the presence of corticosteroids, as assessed and determined by the investigator
* Previously received gene therapy for the treatment of any condition.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) (Dose Escalation Phase) | Baseline to Week 52
  Subjects with at least one TEAE or serious TEAE
Change from baseline in clinical laboratory values (Dose Escalation Phase) | Baseline to Week 52
  Change in serum chemistry values including liver function tests, hematology, and urinalysis
Change from baseline in 12-lead electrocardiograms (ECGs), vital signs, physical examinations (Dose Escalation Phase) | Baseline to Week 52
  Subjects change from baseline in 12-lead electrocardiograms (ECGs), vital signs, physical examinations
Incidence of sustained plasma Phe concentration of ≤360 μmol/L at 28 weeks post dose (Dose Escalation Phase) | Week 28
  Subjects achieving a sustained plasma Phe concentration ≤360 μmol/L at 28 weeks post dose
Change from baseline in Plasma Phe Concentration (Dose Escalation Phase) | Weeks 24-28
  Change from baseline in plasma Phe concentration during Weeks 24-28
Change from baseline in mean Plasma Phe Concentration (Dose Expansion Phase) | Weeks 24-28
  Change from baseline in mean plasma Phe concentration during Weeks 24-28

SECONDARY OUTCOMES:
Incidence of plasma Phe concentration thresholds up to Week 28 post administration of HMI-102 (Dose Expansion Phase) | Baseline to Week 28
  Subjects achieving plasma Phe concentration thresholds up to Week 28 post administration of HMI-102
Incidence of plasma Phe concentration thresholds up to Week 52 post administration of HMI-102 (Dose Expansion Phase) | Baseline to Week 52
  Subjects achieving plasma Phe concentration thresholds up to Week 52 post administration of HMI-102
Change from baseline in total protein intake at Week 52 post-administration of HMI-102 (Dose Expansion Phase) | Week 52
  Subject Achieving a change from baseline in total protein intake at Week 52 post-administration of HMI-102
Incidence and severity of treatment-emergent adverse events (TEAEs) (Dose Expansion Phase) | Baseline to Week 52
  Subjects with at least one TEAE or serious TEAE

OTHER OUTCOMES:
Phenylketonuria Quality of Life Questionnaire (PKU-QOL) | Baseline to Week 52
  Change in PKU-QOL

CONTACTS AND LOCATIONS:
Overall Officials: Olaf A Bodamer, M.D., Principal Investigator — Boston Children's Hospital
Locations (13):
- United States (13):
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - University of South Florida, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The University of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No